CLINICAL TRIAL: NCT01241903
Title: Early Use of Rosuvastatin (Crestor) in Acute Coronary Syndromes: Targeting Platelet-Leukocyte Interactions
Brief Title: Early Use of Rosuvastatin in Acute Coronary Syndromes: Targeting Platelet-Leukocyte Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Susan Smyth (Other)
Responsible Party: Sponsor-Investigator, Susan Smyth, Principal investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-208-F1V
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Acute Coronary Syndrome; Angioplasty, Transluminal, Percutaneous Coronary; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Blood Platelets
Keywords: Platelet activation; platelet leukocyte aggregates
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crestor (Experimental)
  Interventions: Drug: rosuvastatin
- sugar pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rosuvastatin — Patients (n = 54) presenting acute coronary syndrome/non-ST elevation myocardial infarction who present within 8 hours of symptom-onset will be randomized to two groups to receive rosuvastatin (40 mg oral dose) or placebo at the time of presentation, in addition to standard of care (aspirin, clopidogrel, low molecular weight heparin). Blood will be collected at baseline (time of enrollment, immediately prior to drug or placebo), at 6 - 8 hours, at 18 - 24 hours, and at 30 days for analysis of platelet - leukocyte co-aggregate formation, biomarkers of platelet - leukocyte interactions, and biomarkers of myocardial necrosis. Additional samples may be collected just after revascularization, in patients undergoing PCI. The group of patients treated with rosuvastatin will be maintained on rosuvastatin 20 mg daily and the group randomized to placebo will be given rosuvastatin (20 mg oral once daily) within 48 hoursof enrollment and after planned PCI, but before hospital discharge.
  Other Names: crestor
  Arms: Crestor
Drug: placebo — frequency and duration
  Arms: sugar pill

SUMMARY:
The central hypothesis for this work is that platelet - leukocyte interactions play a critical role in the pathogenesis of acute ischemic events. The primary objective of the study is to determine if early, high-dose administration of the HMG-CoA reductase inhibitor rosuvastatin in the setting of acute coronary syndrome and percutaneous coronary intervention exerts beneficial vascular effects by reducing platelet - leukocyte interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 and 80 years old.
2. Subjects must be willing and able to give informed consent
3. A woman of child-bearing potential who is currently sexually active must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for up to 30 days after enrollment.
4. Subjects must have symptoms of acute coronary syndrome as defined by 2 of the 3: (a) history of cardiac-ischemia-related symptoms of at least 10 minutes duration ≤ 8 hours prior to randomized treatment assignment (b) concurrent biomarker evidence of cardiac ischemia, as defined by troponin I or T greater that upper limit of normal (ULN) or creatine kinase-myocardial band (CK-MB) greater than ULN. (c) concurrent electrocardiographic evidence of cardiac ischemia, as defined by new of presumably new ST-segment depression (≥1 mm) or transient (<30 min) ST-segment elevation (≥ 1mm) in at least two contiguous leads.
5. Subjects must be statin naive or currently only on low dose statin (Simvastatin 20mg, Pravastatin 40mg, or Atorvastatin 10mg)

Exclusion Criteria:

* Age <18 years
* Age > 80 years
* Use of Crestor in the past 30 days
* GFR (estimated) <30 ml/min
* Hemodialysis
* History of liver failure
* Unexplained liver function abnormalities
* Current or planned use of cyclosporine or gemfibrozil
* Sepsis
* Hypotension
* Dehydration
* Trauma
* Severe metabolic, endocrine or electrolyte abnormality
* Recent (within the last 2 weeks) or planned (in the next month) major surgery
* HIV/AIDS with current of planned use of HIV protease inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Smyth, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Dept of Cardiology, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects randomized to the placebo arm received a placebo dose at enrollment (day 1) and rosuvastatin 20mg for the next 30 days starting on day 2.
- Rosuvastatin: Subjects randomized to the rosuvastatin arm received rosuvastatin 40mg following enrollment (day 1) and rosustatin 20mg for the next 30 days starting at day 2.
Period: Overall Study
Arm/Group | Placebo | Rosuvastatin
Started | 27 | 27
Completed | 26 | 27
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rosuvastatin | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.7) | 57.2 (10.4) | 56.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet - Leukocyte Aggregates
Description: measured by flow cytometry
Time Frame: within first 24 hours
Measure: Mean (Standard Error); unit: % leukocytes with platelets attached
Arm/Group | Placebo | Rosuvastatin
Number analyzed (Participants) | 24 | 23
% leukocytes with platelets attached
  Baseline | 29.2 (3.8) | 39.8 (4.9)
  8 Hour | 26.2 (4.2) | 21.1 (3.2)
  24 Hour | 24.4 (4.2) | 21.3 (2.8)

2. Secondary Outcome: Biomarkers of Platelet Function and Myocardial Necrosis
Time Frame: up to 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 2/26 | 1/27
Other Adverse Events (participants affected / at risk) | 2/26 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Rosuvastatin (N=27)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject had urine myoglobin 4 hours after randomization. Study drug was discontinued immediately. Symptoms resolved within 40 hours. No clinical signs of rhabdomyolysis were noted. Event was assessed moderate and possibly related to rosuvastatin.
Death (Cardiac disorders) | 1 (1) | 0 (0) — Subject expired from a coronary event 10 days after enrollment. Subject had history of hypertension and a myocardial infarction the day of enrollment. The event was assessed as unrelated to rosuvastatin treatment and caused by underlying disease.
Stroke (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Subject suffered a stroke (acute left hemiparesis) 12 days after enrolling into the study. The stroke was assessed as Grade 3 (severe) and unrelated to rosuvastatin treatment and caused by underlying disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Rosuvastatin (N=27)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject developed rash 3 days after enrollment. Rash resolved after discontinuation of rosuvastatin. Event was assessed as mild and probably related to rosuvastatin.
Alcohol Toxicity (Social circumstances) | 0 (0) | 1 (1) — Subject experienced alcohol toxicity 12 days following enrollment. The event was accessed as mild and probably not related to rosuvastatin.
Nightmare (Social circumstances) | 1 (1) | 0 (0) — Subject complained of experiencing nightmares and flashbacks 14 days after enrollment. Rosuvastatin was discontinued and nightmares continued. The event was assessed as mild and unrelated to rosuvastatin treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No